CLINICAL TRIAL: NCT06749600
Title: Clinical Management and Outcomes of Primary Ovarian Leiomyosarcoma
Acronym: POLMS
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 36/2024/OSS/AUSLRE
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-01

CONDITIONS: Primary Ovarian Leiomyosarcoma
Keywords: Primary ovarian leiomyosarcoma; Gynecologic oncology; Neoplasms, Muscle Tissue; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Sarcoma; Neoplasms; Histopathology; Prognostic factors; Tumor markers
MeSH Terms: conditions — Neoplasms, Muscle Tissue; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Sarcoma; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primary leiomyosarcoma of the ovary (POLMS): The study population includes patients aged between 18 and 99 years diagnosed with primary ovarian leiomyosarcoma (POLMS) afferent to participating centers. This population encompasses both historical cases diagnosed since 1980 and new cases identified during the study period.

SUMMARY:
This observational study aims to gather comprehensive data on primary ovarian leiomyosarcoma (POLMS). This extremely rare malignancy accounts for less than 3% of primary ovarian malignancies and has an incidence of only 1% among ovarian cancers. This national, retrospective and prospective multicenter study will collect and analyze historical cases of POLMS with remote diagnoses accessed through clinical case reviews and newly identified cases. The study aims to expand a previously identified series of 113 cases described in the literature, uncovering patterns in diagnosis, treatment, and outcomes and ultimately establishing evidence-based guidelines for the optimal management of this rare and aggressive cancer.

DETAILED DESCRIPTION:
This study adopts a national, multicenter, observational design, incorporating both retrospective and prospective methodologies to collect and analyze primary ovarian leiomyosarcoma (POLMS) cases. The retrospective component will include cases diagnosed since 1980, leveraging institutional archives and clinical case reviews.

Data collection will be standardized using an electronic Case Report Form (eCRF) implemented on REDCap. All data will be centralized for uniformity and undergo rigorous validation to ensure consistency across centers. Findings will be reported in aggregated form to preserve patient confidentiality.

The study will gather extensive data points, including:

* Patient demographics.
* Clinical presentation and tumor characteristics (symptoms, tumor markers such as CA-125, CEA, and Ki-67).
* Treatment modalities (surgical details, lymphadenectomy, chemotherapy, radiotherapy, or hormonal therapy).
* Recurrence patterns and outcomes (disease-free survival, overall survival).
* Immunohistochemical findings (positivity for desmin, SMA, and vimentin). The statistical analysis primarily involves descriptive and exploratory techniques to identify patterns and correlations within the dataset.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary leiomyosarcoma of the ovary;
* Patients diagnosed with POLMS for whom data relating to diagnosis and treatment are available.
* Aged between 18 and 99 years

Exclusion Criteria:

- All patients with other forms of ovarian sarcoma (rhabdomyosarcomas, fibrosarcomas, stromal cell sarcomas) and patients diagnosed with leiomyosarcoma of the uterus will be excluded.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals assigned female at birth are eligible to participate in this study.
Study Population: Consent for study participation will be obtained from living patients during follow-up visits. Historical cases with remote diagnoses since 1980 will be accessed through clinical case reviews in the databases of each participating center. For patients lost to follow-up or deceased, a waiver of informed consent has been obtained from the Ethics Committee by applicable regulations.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the primary ovarian leiomyosarcoma treatment and prognosis | 3 years observation period
  Correlation between survival outcomes and treatments (type of surgery ,type of chemotherapy, hormone therapy, radiotherapy).

OTHER OUTCOMES:
Correlation between the mitotic index and Ki67 | through study completion, an average of 1 year
  Number of mitotic figures and levels of Ki67 expression in immunohistochemical staining
Correlation between the mitotic index and progression of disease | 3 years observation period
  Correlation between survival outcomes and mitotic index
Overall Survival | 3 years observation period
  Time from diagnosis to death from any cause, measured in months.
Progression free survival in the overall population | 3 years observation period
  Time from diagnosis to disease progression or death, whichever occurs first, measured in months.

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (10):
  - AOU Policlinico di Modena, Modena, Italy
  - Azienda Ospedaliero Universitaria di Parma - S.C. Ostetricia e Ginecologia, Parma, PR
  - Azienda USL IRCCS di Reggio Emilia, Reggio Emilia, RE
  - Malzoni - Avellino, Avellino
  - Azienda Ospedaliero Universitaria Policlinico "G.Rodolico - San Marco" - Catania, Catania
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione Irccs San Gerardo Dei Tintori, Monza
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - Università degli Studi di Napoli Federico II, Napoli
  - Ospedale "Sacro Cuore", Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mandato VD, Torricelli F, Mastrofilippo V, Palicelli A, Costagliola L, Aguzzoli L. Primary Ovarian Leiomyosarcoma Is a Very Rare Entity: A Narrative Review of the Literature. Cancers (Basel). 2023 May 28;15(11):2953. doi: 10.3390/cancers15112953. PMID 37296915
- [Background] Pu T, Fan L, Wang L, Li L, Zeng H. Recurrent primary ovarian leiomyosarcoma preconception, pregnancy, delivery, and puerperal management: A case report and literature review. J Obstet Gynaecol Res. 2022 Jun;48(6):1489-1494. doi: 10.1111/jog.15244. Epub 2022 Mar 30. PMID 35354221
- [Background] Yuksel D, Cakir C, Kilic C, Karalok A, Kimyon G, Coteli S, Boyraz G, Tekin OM, Turan T. Primary leiomyosarcoma of the ovary: a report of three cases and a systematic review of literature. J Gynecol Obstet Hum Reprod. 2021 Jun;50(6):101825. doi: 10.1016/j.jogoh.2020.101825. Epub 2020 Jun 1. PMID 32497729
- [Background] Pongsuvareeyakul T, Sukpan K, Chaicharoen S, Khunamornpong S. Leiomyosarcoma and Squamous Cell Carcinoma Arising in Mature Cystic Teratoma of the Ovary. Case Rep Pathol. 2017;2017:7907359. doi: 10.1155/2017/7907359. Epub 2017 Jul 2. PMID 28751996
- [Background] He M, Deng YJ, Zhao DY, Zhang Y, Wu T. Synchronous leiomyosarcoma and fibroma in a single ovary: A case report and review of the literature. Oncol Lett. 2016 Apr;11(4):2510-2514. doi: 10.3892/ol.2016.4241. Epub 2016 Feb 17. PMID 27073508
- [Background] Zygouris D, Androutsopoulos G, Grigoriadis C, Arnogiannaki N, Terzakis E. Primary ovarian leiomyosarcoma. Eur J Gynaecol Oncol. 2012;33(3):331-3. PMID 22873115
- [Background] Chang A, Schuetze SM, Conrad EU 3rd, Swisshelm KL, Norwood TH, Rubin BP. So-called "inflammatory leiomyosarcoma'': a series of 3 cases providing additional insights into a rare entity. Int J Surg Pathol. 2005 Apr;13(2):185-95. doi: 10.1177/106689690501300210. PMID 15864383
- [Background] Nicotina PA, Antico F, Caruso C, Triolo O. Primary ovarian leiomyosarcoma. Proliferation rate and survival. Eur J Gynaecol Oncol. 2004;25(4):515-6. PMID 15285319
- [Background] Mayerhofer K, Lozanov P, Bodner K, Bodner-Adler B, Mayerhofer-Gallenbacher N, Hudelist G, Czerwenka K. Immunohistochemical analysis of a primary ovarian leiomyosarcoma. Case report. Anticancer Res. 2003 Jul-Aug;23(4):3433-6. PMID 12926085
- [Background] Seracchioli R, Colombo FM, Bagnoli A, Trengia V, Venturoli S. Primary ovarian leiomyosarcoma as a new component in the nevoid basal cell carcinoma syndrome: a case report. Am J Obstet Gynecol. 2003 Apr;188(4):1093-5. doi: 10.1067/mob.2003.86. PMID 12712116
- [Background] Balaton A, Vaury P, Imbert MC, Mussy MA. Primary leiomyosarcoma of the ovary: a histological and immunocytochemical study. Gynecol Oncol. 1987 Sep;28(1):116-20. doi: 10.1016/s0090-8258(87)80016-1. PMID 3308653
- [Background] Nogales FF, Ayala A, Ruiz-Avila I, Sirvent JJ. Myxoid leiomyosarcoma of the ovary: analysis of three cases. Hum Pathol. 1991 Dec;22(12):1268-73. doi: 10.1016/0046-8177(91)90110-b. PMID 1748433
- [Background] Anderson B, Turner DA, Benda J. Ovarian sarcoma. Gynecol Oncol. 1987 Feb;26(2):183-92. doi: 10.1016/0090-8258(87)90272-1. PMID 3643159
- [Background] Shakfeh SM, Woodruff JD. Primary ovarian sarcomas: report of 46 cases and review of the literature. Obstet Gynecol Surv. 1987 Jun;42(6):331-49. No abstract available. PMID 3299172
- [Background] Azoury RS, Woodruff JD. Primary ovarian sarcomas. Report of 43 cases from the Emil Novak Ovarian Tumor Registry. Obstet Gynecol. 1971 Jun;37(6):920-41. No abstract available. PMID 4378308
- [Background] Nieminen U, Numers CV, Purola E. Primary sarcoma of the ovary. Acta Obstet Gynecol Scand. 1969;48(3):423-32. doi: 10.3109/00016346909156657. No abstract available. PMID 5370781
- [Background] KELLEY RR, SCULLY RE. Cancer developing in dermoid cysts of the ovary. A report of 8 cases, including a carcinoid and a leiomyosarcoma. Cancer. 1961 Sep-Oct;14:989-1000. doi: 10.1002/1097-0142(196109/10)14:53.0.co;2-u. No abstract available. PMID 13752348
- [Background] Shafiee MN, Kah Teik C, Md Zain RR, Kampan N. Ovarian and uterine leiomyosarcoma: which one is the primary? Horm Mol Biol Clin Investig. 2019 Aug 9;41(2). doi: 10.1515/hmbci-2019-0037. PMID 31398145
- [Background] Rampaul RS, Barrow S, Naraynsingh V. A primary ovarian leiomyosarcoma with micro-invasive features (stage I): is surgical excision enough? Gynecol Oncol. 1999 Jun;73(3):464; author reply 465-7. doi: 10.1006/gyno.1999.5384. No abstract available. PMID 10366481
- [Background] Dixit S, Singhal S, Baboo HA, Vyas RK, Neema JP, Murthy R, Sooryanaraya U. Leiomyosarcoma of the ovary. J Postgrad Med. 1993 Jul-Sep;39(3):151-3. PMID 8051647
- [Background] Inoue J, Gomibuchi H, Minoura S. A case of a primary ovarian leiomyosarcoma. J Obstet Gynaecol Res. 2000 Dec;26(6):401-7. doi: 10.1111/j.1447-0756.2000.tb01349.x. PMID 11152324
- [Background] Walts AE, Lichtenstein I. Primary leiomyosarcoma associated with serous cystadenocarcinoma of the ovary. Gynecol Oncol. 1977 Mar;5(1):81-6. doi: 10.1016/0090-8258(77)90010-5. No abstract available. PMID 858555
- [Background] Taskin S, Taskin EA, Uzum N, Ataoglu O, Ortac F. Primary ovarian leiomyosarcoma: a review of the clinical and immunohistochemical features of the rare tumor. Obstet Gynecol Surv. 2007 Jul;62(7):480-6. doi: 10.1097/01.ogx.0000268629.16151.71. PMID 17572920
- [Background] Lastarria D, Sachdev RK, Babury RA, Yu HM, Nuovo GJ. Immunohistochemical analysis for desmin in normal and neoplastic ovarian stromal tissue. Arch Pathol Lab Med. 1990 May;114(5):502-5. PMID 2159271
- [Background] Lerwill MF, Sung R, Oliva E, Prat J, Young RH. Smooth muscle tumors of the ovary: a clinicopathologic study of 54 cases emphasizing prognostic criteria, histologic variants, and differential diagnosis. Am J Surg Pathol. 2004 Nov;28(11):1436-51. doi: 10.1097/01.pas.0000141393.99300.d0. PMID 15489647
- [Background] Bouie SM, Cracchiolo B, Heller D. Epithelioid leiomyosarcoma of the ovary. Gynecol Oncol. 2005 May;97(2):697-9. doi: 10.1016/j.ygyno.2005.02.008. PMID 15863185
- [Background] Vijaya Kumar J, Khurana A, Kaur P, Chuahan AK, Singh S. A rare presentation of primary leiomyosarcoma of ovary in a young woman. Ecancermedicalscience. 2015 Apr 21;9:524. doi: 10.3332/ecancer.2015.524. eCollection 2015. PMID 25932048
- [Background] Furutake Y, Fukagawa T, Suga Y, Nagasawa T, Sato S, Omi H, Kagabu M, Chiba A, Shoji T, Takeuchi S, Sugai T, Itamochi H, Sugiyama T. Gemcitabine and docetaxel in a patient with primary ovarian leiomyosarcoma: a case report and review of literature. Int Cancer Conf J. 2017 Sep 11;7(1):11-15. doi: 10.1007/s13691-017-0309-7. eCollection 2018 Jan. PMID 31149505
- [Background] Rasmussen CC, Skilling JS, Sorosky JI, Lager DJ, Buller RE. Stage IIIC ovarian leiomyosarcoma in a premenopausal woman with multiple recurrences: prolonged survival with surgical therapy. Gynecol Oncol. 1997 Sep;66(3):519-25. doi: 10.1006/gyno.1997.4824. PMID 9299270
- [Background] Friedman HD, Mazur MT. Primary ovarian leiomyosarcoma. An immunohistochemical and ultrastructural study. Arch Pathol Lab Med. 1991 Sep;115(9):941-5. PMID 1929791
- [Background] Cojocaru E, Palahepitiva Gamage G, Butler J, Barton DP, Thway K, Fisher C, Messiou C, Miah AB, Zaidi S, Gennatas S, Benson C, Huang P, Jones RL. Clinical management and outcomes of primary ovarian leiomyosarcoma - Experience from a sarcoma specialist unit. Gynecol Oncol Rep. 2021 Mar 2;36:100737. doi: 10.1016/j.gore.2021.100737. eCollection 2021 May. PMID 33732852
- [Background] Monk BJ, Nieberg R, Berek JS. Primary leiomyosarcoma of the ovary in a perimenarchal female. Gynecol Oncol. 1993 Mar;48(3):389-93. doi: 10.1006/gyno.1993.1067. PMID 8462904
- [Background] Arslan OS, Sumer C, Cihangiroglu G, Kanat-Pektas M, Gungor T. A rare tumor of the female genital tract: primary ovarian leiomyosarcoma. Arch Gynecol Obstet. 2011 Mar;283 Suppl 1:83-5. doi: 10.1007/s00404-010-1735-3. PMID 21061129
- [Background] Goodall EJ, Madhuri T, Manuel SB. The Management Dilemma of Leiomyosarcoma of the Ovary. World J Oncol. 2011 Oct;2(5):265-266. doi: 10.4021/wjon362w. Epub 2011 Oct 28. PMID 29147259
- [Background] Pankaj, S., Choudhary, V., Singh, R. K., & Harsvardhan, R. (2013). High grade pleomorphic leiomyosarcoma of ovary in a young female: a case report. World Journal of Surgical Research, 2(3).